CLINICAL TRIAL: NCT03122067
Title: Oxytocinergic Modulation of Perceived Social Exclusion
Brief Title: Oxytocin's Effect on Social Pain Empathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-33
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: oxytocin; social cognition; fMRI; empathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin group (Experimental): male participants with oxytocin treatment
  Interventions: Drug: oxytocin treatment
- placebo group (Placebo Comparator): male participants with placebo treatment
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: oxytocin treatment — intranasal administration of oxytocin
  Arms: oxytocin group
Drug: placebo treatment — intranasal administration of placebo
  Arms: placebo group

SUMMARY:
The aim of the present experiment is to examine oxytocin's behavioral and neural effects on social pain empathy

DETAILED DESCRIPTION:
In the current study, the investigators plan to examine whether oxytocin modulates behavior and neural activity during observing another person being excluded in an online ball-tossing game (a modified cyberball paradigm).

ELIGIBILITY:
Inclusion Criteria:

* healthy participants without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness
* smoking or drinking 24 hours before experiment

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Neural activity changes associated with oxytocin administration | 45-60 minutes after drug administration
  fMRI-assessed brain activity during observing other being socially excluded

SECONDARY OUTCOMES:
Behavioral changes associated with oxytocin administration: ball-tossing | 45-60 minutes after drug administration
  Number of tosses to the other players (the excluder, new player, or previously excluded player)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China